CLINICAL TRIAL: NCT03130127
Title: Continuous Versus Bolus Infusion of Terlipressin for Portal Hypertension Related Bleeding in Liver Cirrhosis: A Prospective Non-randomized Controlled Trial
Brief Title: Continuous Versus Bolus Infusion of Terlipressin for Portal Hypertension Related Bleeding in Liver Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Doctor, General Hospital of Shenyang Military Region
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERLIPRESSIN-LC
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Variceal Hemorrhage; Bleeding; Esophageal and Gastric Varices
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Hemorrhage; Esophageal and Gastric Varices | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous infusion of terlipressin (Experimental): In our clinical practice, continuous infusion of terlipressin is being employed.
  Interventions: Drug: Terlipressin
- Bolus infusion of terlipressin (Active Comparator): Traditionally, a bolus infusion of terlipressin is recommended.
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — According to the current practice guidelines and consensus, terlipressin is the standard treatment option for acute variceal bleeding in liver cirrhosis.
  Other Names: Glypressin

SUMMARY:
Terlipressin is the mainstay drug for the treatment of acute variceal bleeding in liver cirrhosis. According to the drug instructions, intravenous bolus infusion is the standard approach of terlipressin. It remains unclear about whether or not continuous infusion of terlipressin should be considered.

DETAILED DESCRIPTION:
Although intravenous bolus infusion of terlipressin is the standard approach, continuous infusion of terlipressin is preferred in clinical practice. The present study is a pilot non-randomized controlled trial to explore the feasibility and safety of continuous infusion of terlipressin for the treatment of acute variceal bleeding in liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of liver cirrhosis;
2. Child-Pugh B or C;
3. Acute gastroesophageal variceal bleeding;
4. Written informed consents. -

Exclusion Criteria:

1. No liver cirrhosis;
2. Child-Pugh class A;
3. Acute upper gastrointestinal bleeding unrelated to varices;
4. Use of somatostatin or octreotide. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
5 day treatment failure | 5 days (120 hours)
  Death, fresh hematemesis, hypovolaemic shock, or 3 g drop in Hb (9% drop of Ht) within any 24 h period if no transfusion is administered.

SECONDARY OUTCOMES:
Six-week mortality | 6 weeks
  Death with 6 weeks after treatment

OTHER OUTCOMES:
Adverse events related to terlipressin [Safety] | 5 days after treatment
  Adverse events related to terlipressin, such as hyponatremia, diarrhea, abdominal pain, arterial hypertension, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Guo, MD, Principal Investigator — General Hospital of Shenyang Military Area

IPD SHARING:
Plan to Share IPD: No